CLINICAL TRIAL: NCT00089193
Title: Evaluation of GM-CSF-in-Adjuvant and the Number of Vaccine Sites on Immunization With Multiple Synthetic Melanoma Peptides
Brief Title: Vaccine Therapy With or Without Sargramostim in Treating Patients With Stage IIB, Stage IIC, Stage III, or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Craig L Slingluff, Jr (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Craig L Slingluff, Jr, Professor, Department of Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 10524; UVACC-MEL-43; FCCC-03045; MDA-2003-0720
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Melanoma (Skin)
Keywords: stage II melanoma; stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — incomplete Freund's adjuvant; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: incomplete Freund's adjuvant
Biological: multi-epitope melanoma peptide vaccine
Biological: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Combining vaccine therapy with sargramostim may cause a stronger immune response and kill more tumor cells.

PURPOSE: This randomized phase II trial is studying vaccine therapy and sargramostim to see how well they work compared to vaccine therapy alone in treating patients with stage II B, stage IIC, stage III, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare immune response in patients with stage IIB-IV melanoma treated with vaccination comprising multiple synthetic melanoma peptides and Montanide ISA-51 with vs without sargramostim (GM-CSF).
* Compare immune response in patients treated with these vaccinations administered at 1 vs 2 sites.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive vaccination comprising multiple synthetic melanoma peptides and Montanide ISA-51 at 1 injection site.
* Arm II: Patients receive vaccination comprising multiple synthetic melanoma peptides and Montanide ISA-51 at 2 injection sites.
* Arm III: Patients receive vaccination comprising multiple synthetic melanoma peptides, Montanide ISA-51, and sargramostim (GM-CSF) at 1 injection site.
* Arm IV: Patients receive vaccination comprising multiple synthetic melanoma peptides, Montanide ISA-51, and GM-CSF at 2 injection sites.

In all arms, treatment repeats once weekly for 6 weeks. Patients return for booster vaccinations at weeks 12, 26, 39, and 52.

PROJECTED ACCRUAL: A maximum of 124 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of melanoma

  * Stage IIB, IIC, III, or IV disease
* Must express HLA-A1, -A2, or -A3
* No ocular melanoma

PATIENT CHARACTERISTICS:

Age

* 12 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL

Hepatic

* Liver function tests ≤ 2.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Not pregnant or nursing
* No other malignancy within the past 5 years except basal cell or squamous cell skin cancer without brain metastasis, carcinoma in situ of the breast, or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior growth factors
* More than 4 weeks since prior allergy shots
* No prior vaccine therapy for melanoma or any other cancer with any of the peptides used in this study
* More than 12 weeks since prior melanoma vaccine therapy* NOTE: *Prior melanoma vaccine allowed only for patients with disease progression during or after administration of the vaccine

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior steroids

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-09; Primary Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Study Chair — University of Virginia
Locations (5):
- United States (5):
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center at University of Texas, Houston, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Clancy-Thompson E, King LK, Nunnley LD, Mullins IM, Slingluff CL Jr, Mullins DW. Peptide vaccination in Montanide adjuvant induces and GM-CSF increases CXCR3 and cutaneous lymphocyte antigen expression by tumor antigen-specific CD8 T cells. Cancer Immunol Res. 2013 Nov;1(5):332-9. doi: 10.1158/2326-6066.CIR-13-0084. PMID 24377099